CLINICAL TRIAL: NCT06937593
Title: A Phase 1, Randomized, Placebo-controlled, Double-blind, Multiple Ascending Dose Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VIS954 in Healthy Participants
Brief Title: A Study to Evaluate Safety, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Multiple Doses of VIS954
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Visterra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIS954-102
Record Dates: First submitted 2025-04-09; First posted 2025-04-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VIS954 - Low Dose (Experimental): VIS954 Low Dose will be administered subcutaneously on Days 1, 15, 29, 43, 57, and 71
  Interventions: Drug: VIS954
- VIS954 - Medium Dose (Experimental): VIS954 Medium Dose will be administered subcutaneously on Days 1, 15, 29, 43, 57, and 71
  Interventions: Drug: VIS954
- VIS954 - High Dose (Experimental): VIS954 High Dose will be administered subcutaneously on Days 1, 15, 29, 43, 57, and 71
  Interventions: Drug: VIS954
- Placebo (Placebo Comparator): Placebo will be administered subcutaneously on Days 1, 15, 29, 43, 57, and 71
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIS954 — A humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb)
  Arms: VIS954 - High Dose; VIS954 - Low Dose; VIS954 - Medium Dose
Drug: Placebo — VIS954 Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and pharmacodynamics of multiple doses of VIS954 compared with placebo in healthy adult participants.

DETAILED DESCRIPTION:
The study will be conducted in 3 sequential cohorts. Each cohort will enroll 8 participants, randomized to VIS954 or placebo at a ratio of 6:2.

In each cohort, participants will be administered 6 doses of VIS954 or placebo with a dosing frequency of once every 2 weeks (Q2W). A Safety Monitoring Committee (SMC) will review the data and approve escalation to the next planned dose level.

The total duration of the clinical trial for each participant will be up to approximately 7 months, including the screening period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant between 18 and 55 years of age, inclusive, at the screening visit.
2. Body mass index between 18.0 and 30.0 kg/m2, inclusive, at the screening visit.
3. Total body weight between 50.0 and 120.0 kg, inclusive, at the screening visit.
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
5. Willing and able to participate in the trial for the defined duration of the trial.
6. Female participants will be nonpregnant, nonlactating, and either postmenopausal for at least 1 year or surgically sterile for at least 3 months, or will agree to use highly effective methods of contraception from the period prior to trial enrollment until 90 days after Week 20 (or the last dose); women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) test at screening.
7. Male participants must agree to use double barrier contraception or abstain from sex during the trial and until 90 days after Week 20 (or the last dose). Male participants must agree to refrain from sperm donation for the duration of the trial and until 150 days after the last dose. This criterion may be waived for male participants who have had a vasectomy greater than 6 months prior to enrollment.
8. Healthy, as determined by pretrial medical evaluation (medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests), as judged by the principal investigator.

Exclusion Criteria:

1. Participant has a history or current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, hematologic, autoimmune, blood dyscrasias or other medical disorder, including psychiatric disorders, cirrhosis, or treated, limited cervical carcinomas (ie, carcinoma in situ) are not exclusionary.
2. Participant is participating in another clinical trial of any investigational drug, device, or intervention or has received any investigational medication during the last 30 days or 5 half-lives, whichever is longer, before baseline (Day -1).
3. Previous receipt of antibody or biologic therapy.
4. Receipt of blood products within 6 months prior to screening.
5. History of a previous hypersensitivity or severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis to any of the ingredients of the VIS954 subcutaneous (SC) injection formulation.
6. Previous exposure to VIS954.
7. Blood pressure > 140/90 mmHg or < 90/60 mmHg (may be repeated once if abnormal), at the screening visit or Day -1.
8. History of any infection requiring hospitalization or treatment with antivirals, antibiotics, or systemic antifungals within 3 months prior to screening.
9. Received a vaccination, other than Coronavirus Disease 2019 (COVID-19) vaccination, during the 30 days prior to administration of the first dose of study intervention. A COVID-19 vaccination cannot be received within 7 days prior to the first dose of study intervention and until 14 days after the last dose.
10. Has received any prescription or nonprescription (over-the-counter) medication during the last 30 days or 5 half-lives, whichever is longer, preceding baseline (Day -1), with the exception of acetaminophen, ibuprofen, naproxen (or other over-the-counter nonsteroidal anti-inflammatory drugs [NSAID]), hormonal contraceptives, topical medications, vitamins, and dietary or herbal remedies.
11. Any participant who has a recent history of alcohol or drug/chemical abuse, at the discretion of the investigator, will be excluded.
12. For the duration of the trial, enrolled male participants should not consume more than 15 standard drinks per week (7 days) and female participants should not consume more than 10 standard drinks per week (7 days). A standard drink equals 10 g of alcohol. Enrolled participants must abstain from consuming alcohol 48 hours prior to each administration of study intervention.
13. Enrolled participants must abstain from consumption of nicotine containing products from Day-1 through discharge from the trial site clinic (Day 3).
14. Enrolled participants must abstain from consumption of cannabinoids from Day-1 through end of trial.
15. Participant with a positive urine drug and alcohol screen test result at screening or baseline. The urine drug and alcohol screen may be repeated once at the discretion of the investigator. The urine drug screen includes screening for cannabinoids, methylenedioxymethamphetamine, and propoxyphene. If a participant tests positive on these tests, inclusion of that participant into the trial will be based on the principal investigator's judgment with consultation, as needed, with the medical monitor and the sponsor.
16. Any chronic infectious disease (eg, chronic urinary tract infection, chronic sinusitis, bronchiectasis, active pulmonary or systemic tuberculosis [TB], chronic viral hepatitis such as hepatitis C or hepatitis B, or human immunodeficiency virus [HIV] infection).
17. Participant who has donated > 500 mL of blood within 60 days prior to start of the screening visit or the participant has donated any plasma within 7 days prior to baseline (Day -1).
18. Coronavirus disease 2019 (COVID-19):

    * Current symptoms of infection.
    * Diagnosis of COVID-19 (reverse transcription polymerase chain reaction [RT-PCR], antigen testing, or clinical diagnosis) in the 21 days prior to screening.
    * Ongoing diagnosis of "Long-COVID" symptoms, due to a prior COVID-19 infection.
19. Is an employee of the clinical research team (any sponsor or research site employee), or has a family member who is an employee of these organizations.
20. Participant is judged by the investigator or the medical monitor to be inappropriate for the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 169 days
  Number and Percentage of Adverse Events (AEs) that first occurred or worsened in severity after the study intervention administration.
Maximum serum concentration after administration of VIS954 over time | 169 days
  Blood samples will be collected for measurement of serum concentrations of VIS954 at specified time points to assess maximum serum concentration over time
Area under the concentration-time curve from time zero extrapolated to time t | 169 days
  Blood samples will be collected for measurement of serum concentrations of VIS954 at specified time points to assess area under the concentration-time curve from time zero extrapolated to time t (AUC 0-t)

SECONDARY OUTCOMES:
VIS954 Percentage Receptor Occupancy | 169 days
  Pharmacodynamic parameter to characterize and evaluate VIS954 binding to target receptor

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Winkle, MD, Principal Investigator — Anaheim Clinical Trials
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States